CLINICAL TRIAL: NCT01032967
Title: Multicenter Prospective Randomized Trial Comparing Standard Esophagectomy With Chemoradiotherapy for Treatment of Squamous Esophageal Cancer: Early Results From the Chinese University Research Group for Esophageal Cancer (CURE)
Brief Title: Surgery or Chemoradiation for Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Professor Philip Chiu, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Surgery or CRT Ca Esophagus
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancers
Keywords: squamous cell carcinoma; esophagectomy; chemoradiotherapy; chemoradiation; Squamous cell carcinomas of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery, esophagectomy (Active Comparator): The patients randomized to receive either standard esophagectomy will have the operation performed in an open manner with two-field lymphadenectomy
  Interventions: Procedure: Esophagectomy
- Definitive chemoradiation (Active Comparator): 3-weekly cycles of cisplatin and 5-fluorouracil chemotherapy and radical radiotherapy delivered in a three-dimensional conformal mode (total of 50-60 Gy given in 25-30 fractions) will be given over a period 5-6 weeks.
  Interventions: Radiation: Definitive chemoradiation

INTERVENTIONS:
Procedure: Esophagectomy — The patients will receive standard open esophagectomy with two-field lymphadenectomy
  Arms: Surgery, esophagectomy
Radiation: Definitive chemoradiation — 3-weekly cycles of cisplatin and 5-fluorouracil chemotherapy and radical radiotherapy delivered in a three-dimensional conformal mode (total of 50-60 Gy given in 25-30 fractions) will be given over a period 5-6 weeks.
  Arms: Definitive chemoradiation

SUMMARY:
The aim of this study is to compare outcomes in patients with operable squamous carcinoma of the esophagus who have received either surgery or definitive chemoradiation (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients had mid or lower thoracic esophageal cancers that were confirmed on histology to be a squamous cell carcinoma deemed to be resectable.

Exclusion Criteria:

* The investigators excluded those patients who had distant metastasis to solid visceral organs or local invasion into trachea, descending aorta, or recurrent laryngeal nerve.
* Those patients who were older than 75 years or who had a serious premorbid condition or a poor physical status that compromised a thoracotomy were also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Overall survival and disease-free survival | 2 year and 5 year

SECONDARY OUTCOMES:
Quality of life and function outcomes | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Philip W Chiu, FRCSEd (Gen), Principal Investigator — Chinese University of Hong Kong

REFERENCES:
- [Derived] Teoh AY, Chiu PW, Yeung WK, Liu SY, Wong SK, Ng EK. Long-term survival outcomes after definitive chemoradiation versus surgery in patients with resectable squamous carcinoma of the esophagus: results from a randomized controlled trial. Ann Oncol. 2013 Jan;24(1):165-71. doi: 10.1093/annonc/mds206. Epub 2012 Aug 10. PMID 22887465
- [Derived] Teoh AY, Yan Chiu PW, Wong TC, Liu SY, Hung Wong SK, Ng EK. Functional performance and quality of life in patients with squamous esophageal carcinoma receiving surgery or chemoradiation: results from a randomized trial. Ann Surg. 2011 Jan;253(1):1-5. doi: 10.1097/SLA.0b013e3181fcd991. PMID 21233603